CLINICAL TRIAL: NCT02092324
Title: Prospective Evaluation of Ruxolitinib Efficacy for CNL/aCML Patients With Mutation of CSF3R
Brief Title: Ruxolitinib Phosphate in Treating Patients With Chronic Neutrophilic Leukemia or Atypical Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Kim-Hien Dao, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010262; NCI-2014-00633 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00010262 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Chronic Neutrophilic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Neutrophilic, Chronic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ruxolitinib phosphate) (Experimental): Patients receive ruxolitinib phosphate PO every other day, QD, or BID on days 1-28. Each patient will be followed for a maximum of 96 weeks (24 cycles, 1 cycle is 4 weeks long). If the study drug continues to be effective, the patient may be eligible to continue on study drug past 24 cycles.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase II trial studies how well ruxolitinib phosphate works in treating patients with chronic neutrophilic leukemia (CNL) or atypical chronic myeloid leukemia (aCML). Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cells to reproduce. This trial also studies the genetic makeup of patients. Certain genes in cancer cells may determine how the cancer grows or spreads and how it may respond to different drugs. Studying how the genes associated with CNL and aCML respond to the study drug may help doctors learn more about CNL and aCML and improve the treatment for these diseases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients with chronic neutrophilic leukemia (CNL) and atypical chronic myeloid leukemia (aCML) who have a hematologic response to ruxolitinib (ruxolitinib phosphate) (partial response [PR], complete response [CR], complete response, partial [CRp]).

SECONDARY OBJECTIVES:

I. To determine the frequency of grade 3 or 4 hematologic and non-hematologic adverse events experienced by subjects during therapy with ruxolitinib.

II. To determine whether hematologic responses correlate with certain types of mutations in colony stimulating factor 3 receptor (CSF3R) and reduction in mutant CSF3R allele burden in the peripheral blood.

III. To determine the maximum clinical responses for each subject and the median duration of maximum clinical responses.

IV. To determine the mean % reduction of spleen size, estimated by volume using the conventional prolate ellipsoid method as measured by ultrasound compare to baseline.

V. To determine the mean % reduction of total symptom score as measured by a modified Myeloproliferative Neoplasm Symptom Assessment Form version 2.0 (MPN-SAF) compared to start of study (day 1, cycle 1).

VI. To determine overall survival in subjects who complete a minimum of 1 dose of study drug.

VII. To determine the proportion of subjects who discontinue after completion of > 3 cycles but < 6 cycles.

VIII. To determine the proportion of subjects who discontinue prior to completion of cycle 3.

OUTLINE:

Patients receive ruxolitinib phosphate orally (PO) every other day, once daily (QD), or twice daily (BID) on days 1-28. Each patient will be followed for a maximum of 96 weeks (24 cycles, 1 cycle is 4 weeks long). If the study drug continues to be effective, the patient may be eligible to continue on study drug past 24 cycles.

After completion of study treatment, patients are followed up within 2 weeks and at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be newly diagnosed or previously diagnosed with CNL or aCML; all patients must have a bone marrow biopsy completed during the screening or baseline period if one has not been done within 90 days of day 1, cycle one
* Subjects must have platelet count greater than 25,000 per microliter at baseline and at the start of study (day 1, cycle 1) visit
* Subjects must be able to discontinue any drug treatment aimed at lowering disease burden in CNL or aCML; subjects should discontinue hydroxyurea to treat underlying CNL or aCML disease no later than day -7 (one week before starting ruxolitinib); for drugs that have more long-lasting effects on the marrow, such as thalidomide and its analogs, and interferon, subjects should discontinue these no later than day -28
* Subjects must be willing to accept/continue transfusions to treat low hemoglobin levels
* Subjects must have a life expectancy of > 6 months

Exclusion Criteria:

* Subjects unable to review and sign informed consent form
* Females who are pregnant or breastfeeding, and males and females who cannot comply with requirements to avoid fathering a child or becoming pregnant
* Subjects with known diagnosis of human immunodeficiency virus (HIV) or chronic active Hepatitis B or C; viral testing is not required; subjects with a history of Hepatitis B and/or C are allowed on trial if the virus is undetected at the time of enrollment
* Subjects with inadequate liver (alanine aminotransferase [ALT]/serum glutamate pyruvate transaminase [SGPT] above 4 X upper limit of normal [ULN] or direct bilirubin 4 X ULN AND the lab abnormalities are felt to be due to underlying liver dysfunction)
* Subjects with end stage renal function (creatinine clearance [CrCl] < 15 mL/min or glomerular filtration rate [GFR] <15 mL/min) regardless of whether hemodialysis is required
* Subjects with clinically serious infections requiring ongoing antibiotic therapy
* Subjects with severe (immediately life threatening) and recent (occurring within the last 3 months) cardiac dysfunction, pulmonary dysfunction, esophageal variceal bleeding, hemorrhagic strokes, or intracranial hemorrhage are not eligible for study participation
* Subjects requiring therapeutic doses of anticoagulation or anti-platelet therapies (aspirin above 81 mg daily, Plavix or similar agents) AND platelet counts are below 50,000 on two different laboratory evaluations, separated by minimum of two weeks
* Taking investigational or commercial agents or therapies with the intent to treat the subject's malignancy other than those therapies permitted
* Subjects with invasive malignancy over the previous 2 years except treated early stage carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, and completely resected papillary thyroid and follicular thyroid cancers
* Previous allergic reactions to janus kinase (JAK) inhibitors or excipients
* Prior therapy with ruxolitinib or other JAK inhibitors
* Subjects who have had major surgery within 4 weeks prior to entering the study
* Subjects who are anticipated to receive a transplant within the first 6 months of treatment on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim-Hien Dao, Principal Investigator — OHSU Knight Cancer Institute
Locations (7):
- United States (7):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Savona MR, Malcovati L, Komrokji R, Tiu RV, Mughal TI, Orazi A, Kiladjian JJ, Padron E, Solary E, Tibes R, Itzykson R, Cazzola M, Mesa R, Maciejewski J, Fenaux P, Garcia-Manero G, Gerds A, Sanz G, Niemeyer CM, Cervantes F, Germing U, Cross NC, List AF; MDS/MPN International Working Group. An international consortium proposal of uniform response criteria for myelodysplastic/myeloproliferative neoplasms (MDS/MPN) in adults. Blood. 2015 Mar 19;125(12):1857-65. doi: 10.1182/blood-2014-10-607341. Epub 2015 Jan 26. PMID 25624319
- [Result] Dao KT, Gotlib J, Deininger MMN, Oh ST, Cortes JE, Collins RH Jr, Winton EF, Parker DR, Lee H, Reister A, Schultz, Savage S, Stevens, Brockett C, Subbiah N, Press RD, Raess PW, Cascio M, Dunlap J, Chen Y, Degnin C, Maxson JE, Tognon CE, Macey T, Druker BJ, Tyner JW. Efficacy of Ruxolitinib in Patients With Chronic Neutrophilic Leukemia and Atypical Chronic Myeloid Leukemia. J Clin Oncol. 2020 Apr 1;38(10):1006-1018. doi: 10.1200/JCO.19.00895. Epub 2019 Dec 27. PMID 31880950
- [Derived] Dao KH, Solti MB, Maxson JE, Winton EF, Press RD, Druker BJ, Tyner JW. Significant clinical response to JAK1/2 inhibition in a patient with CSF3R-T618I-positive atypical chronic myeloid leukemia. Leuk Res Rep. 2014 Aug 1;3(2):67-9. doi: 10.1016/j.lrr.2014.07.002. eCollection 2014. PMID 25180155
- See also: An international consortium proposal of uniform response criteria for myelodysplastic/myeloprolierative neoplasms (MDS/MPN) in adults — https://pubmed.ncbi.nlm.nih.gov/25624319/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled July 8, 2014 and recruitment ended in September 2019, across seven medical centers in the US.
Pre-assignment Details: Two subjects who were enrolled were shortly determined to be misdiagnosed and were not evaluable bringing the total eligible subjects to 49. An additional subject was not evaluable for the primary endpoint because of missing bone marrow (BM) biopsy data.
Groups:
- Treatment (Ruxolitinib Phosphate): Patients receive ruxolitinib phosphate PO every other day (QOD), or twice a day (BID) on days 1-28. Each patient will be followed for a maximum of 96 weeks (24 cycles, 1 cycle is 4 weeks long). If the study drug continues to be effective, the patient may be eligible to continue on study drug past 24 cycles.
Period: Overall Study
Arm/Group | Treatment (Ruxolitinib Phosphate)
Started | 51
End of Cycle 6 (We expanded accrual to enroll additional evaluable subjects for analysis of the secondary endpoints.) | 25 (This study has an accrual goal of 25 evaluable subjects who reach cycle 7, week 1.)
Wildtype CSF3R (Participants were stratified by CSF3R mutation status) | 23
Mutant CSF3R (Participants were stratified by CSF3R mutation status) | 26
Completed | 32
Not Completed | 19
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 6
Not completed — Proceed to Transplant | 3
Not completed — Physician Decision | 7
Not completed — Misdiagnosis | 2

BASELINE CHARACTERISTICS:
Groups:
- Wildtype CSF3R: Subjects with wild type granulocyte Colony Stimulating Factor Receptor 3 (CSF3R)
- Mutant CSF3R: Subjects with mutant CSF3R
- Total: Total of all reporting groups
Arm/Group | Wildtype CSF3R | Mutant CSF3R | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Median (Full Range); unit: years] | 72.8 [43.1 to 90.7] | 73.0 [60.2 to 92.3] | 72.8 [43.1 to 92.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 26 | 47
  Black or African American | 2 | 0 | 2
Disease group [Count of Participants; unit: Participants]
  CNL | 5 | 17 | 22
  aCML | 18 | 9 | 27
Splenomegaly at baseline [Count of Participants; unit: Participants]
  No Splenomegaly | 6 | 3 | 9
  Splenomegaly | 17 | 23 | 40
Spleen volume by ultrasound [Median (Full Range); unit: cm^3] — Population: Four subjects did not have baseline spleen size evaluated in three-dimensions by ultrasound
  cm^3
    number analyzed (Participants) | 20 | 25 | 45
    (all) | 582.8 [147.4 to 3042.4] | 586.9 [96.2 to 2578.6] | 586.9 [96.2 to 3042.4]
Palpable spleen length at left midcostochondral line (LMC) [Median (Full Range); unit: cm] — Population: 17 subjects did not have measureable or palpable spleen at baseline
  cm
    number analyzed (Participants) | 15 | 17 | 32
    (all) | 9.0 [0.0 to 26.0] | 5.0 [0.0 to 18.0] | 5.8 [0.0 to 26.0]
White blood cell count [Median (Full Range); unit: 10^9 cells/L] | 48.1 [8.5 to 256.9] | 51.6 [6.6 to 209.0] | 50.7 [6.6 to 256.9]
Absolute Neutrophil Count (ANC) [Median (Full Range); unit: 10^9 cells/L] | 35.4 [6.9 to 105.3] | 46.0 [6.1 to 200.6] | 41.9 [6.1 to 200.6]
Hemoglobin [Median (Full Range); unit: g/dL] | 11.0 [7.0 to 14.5] | 10.4 [6.7 to 13.3] | 10.8 [6.7 to 14.5]
Platelets [Median (Full Range); unit: 10^9 cells/L] | 134 [25 to 488] | 125 [26 to 423] | 130 [25 to 488]
Prior therapy [Count of Participants; unit: Participants]
  None | 10 | 8 | 18
  Prior therapy | 13 | 18 | 31
Type of prior therapy [Count of Participants; unit: Participants]
  Hydroxyurea | 11 | 15 | 26
  Hydroxyurea + Azacitidine | 1 | 0 | 1
  Hydroxyurea + Dasatinib | 1 | 0 | 1
  Decitabine | 0 | 2 | 2
  Other (interferon) | 0 | 1 | 1
  No prior treatment | 10 | 8 | 18
IPSS total score [Median (Full Range); unit: units on a scale] — International Prognostic Scoring System (IPSS), based on three prognostic indicators, with values ranging from 0 - 5 where 0 indicates "Low Risk"; 1 indicates "Intermediate 1 Risk"; 2 indicates "Intermediate 2 Risk"; 3 and above indicate "High Risk".
  units on a scale | 2.0 [1.0 to 5.0] | 2.5 [1.0 to 5.0] | 2.0 [1.0 to 5.0]
MPN-SAF TSS [Median (Full Range); unit: units on a scale] — Myeloproliferative Neoplasm Symptom Assessment Form Total symptom score (MPN-SAF TSS) ranges from 0 (no symptoms) to 10 (worst imaginable symptoms). The score is a composite of 10 independent measurements, generating a final score ranging from 0 - 100. Although lower scores indicate fewer symptoms, not all symptoms directly relate to outcomes. Population: Three subjects failed to respond to all 10 questions required to score TSS
  units on a scale
    number analyzed (Participants) | 21 | 25 | 46
    (all) | 28.0 [0.0 to 72.0] | 20.0 [2.0 to 53.0] | 23.5 [0.0 to 72.0]
Prestudy disease duration, months [Median (Full Range); unit: months] | 0.9 [0.2 to 24.9] | 1.2 [0.0 to 64.1] | 0.9 [0.0 to 64.1]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of First 25 Enrolled Patients With a Hematologic Response to Ruxolitinib (Complete Response (CR), Partial Response (PR))
Description: A subject is defined as being responsive (responder) if he or she has achieved complete response (CR) or partial response (PR) at the beginning of cycle 7 compared to start of study (day 1,cycle 1). Subjects who do not reach the start of cycle 7 are counted as non-responders. Proportions with 95% exact confidence intervals will be computed. Protocol-defined Response evaluates changes in white blood cell count, absolute neutrophil count, marrow findings and spleen size to define response (attached protocol, Section 10.6, Clinical Response, Table 6 and Table). IWG-defined Response evaluates bone marrow cellularity and myeloblast percent, absence of osteopmyelofibrosis, peripheral blood elements (white blood cell, Neutrophil, Monocyte and platelet counts, hemoglobin density, percent blasts and Neutrophil precursors), symptom resolution, dysplasia, and spleen size to determine response (attached reference).
Time Frame: Start of cycle 7
Population: First 25 enrolled subjects enrolled, received at least one dose of study drug, and were evaluated for protocol-defined and International Working Group (IWG) defined objective response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- First 25 Enrolled Subjects: First 25 enrolled subjects evaluated for protocol-defined objective response
Arm/Group | First 25 Enrolled Subjects
Number analyzed (Participants) | 25
percentage of participants
  Protocol-defined Response | 32 [15 to 54]
  IWG-defined Response | 4 [0.1 to 20]
Statistical Analysis 1: Comparison: First 25 Enrolled Subjects; Proportion estimated using Clopper-Pearson method. P-value is one-sided proportion test for greater than 10% response rate (based on Simon's 2-stage); Test type: Superiority — 1-proportion test for greater than 10% difference; p = 0.002, binomial — p-value for Protocol-defined objective response
Statistical Analysis 2: Comparison: First 25 Enrolled Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — 1-proportion test for greater than 10% difference; p = 0.90, binomial — p-value is for IWG-defined objective response

2. Secondary Outcome: Percentage of Participant With Any Hematologic Grade III or IV Adverse Events.
Description: The frequency (percentage) of subjects with any hematologic [thrombocytopenia, anemia or neutropenia] grade III or IV adverse events according to CTCAE v4.0
Time Frame: Up to 6 weeks after last dose of ruxolitinib phosphate
Population: All subjects receiving at least one dose of ruxolitinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants | 46.9 [32.5 to 61.7]

3. Secondary Outcome: Percentage of Participants With Any Non-hematologic Grade III or IV Adverse Events.
Description: The frequency (percentage) of subjects with any non-hematologic grade III or IV adverse events according to CTCAE v4.0
Time Frame: Up to 6 weeks after last dose of ruxolitinib phosphate
Population: All subjects receiving at least one dose of ruxolitinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants | 69.4 [54.6 to 81.7]

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response of Partial Response or Better
Description: Compute the percent of patients with protocol-defined objective response (CR+PR) and IWG-defined objective response (CR+PR) at the start of cycle 7 among all enrolled patients (n = 49). Patients who withdrew prior to the end of cycle 6 are considered non-responders. Protocol-defined Response evaluates changes in white blood cell count, absolute neutrophil count, marrow findings and spleen size to define response (attached protocol, Section 10.6, Clinical Response, Table 6 and Table). IWG-defined Response evaluates bone marrow cellularity and myeloblast percent, absence of osteopmyelofibrosis, peripheral blood elements (white blood cell, Neutrophil, Monocyte and platelet counts, hemoglobin density, percent blasts and Neutrophil precursors), symptom resolution, dysplasia, and spleen size to determine response (attached reference).
Time Frame: Start of cycle 7
Population: All enrolled subjects who receive at least one dose of ruxolitinib. Subjects who withdraw prior to the start of cycle 7 are considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants
  Protocol-defined Response | 33 [20 to 48]
  IWG-defined Response | 8 [2.3 to 20]
Statistical Analysis 1: Comparison: Treatment (Ruxolitinib Phosphate); Test type: Superiority — Proportion estimated using Clopper-Pearson method. P-value is one-sided proportion test for greater than 10% response rate; p < 0.0001, Clopper-Pearson method — p-value for protocol-defined objective response. p-value for IWG-defined objective response is 0.70
Statistical Analysis 2: Comparison: Treatment (Ruxolitinib Phosphate); Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.70, Clopper-Pearson method — p-value for IWG-defined objective response

5. Secondary Outcome: Median Time on Study (Months) for Early Drop Offs
Description: Median and range of months on study for subjects who did not complete 6 cycles of Ruxolitinib
Time Frame: End of cycle 6
Population: Enrolled subjects who received at least one dose of study drug but did not complete 6 full cycles of Ruxolitinib
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 17
months | 2.4 [.2 to 5.7]

6. Secondary Outcome: Median Time on Study (Months) for All Enrolled Subjects
Description: Median and range of months on Ruxolitinib for all enrolled subjects
Time Frame: Outcome is measured from the first dose of study drug. If study drug continues to be effective, patient may be eligible to continue on study drug past 24 cycles (up to 4.5 years)
Population: Enrolled subjects who received at least one dose of Ruxolitinib
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
months | 8.5 [.2 to 50.5]

7. Secondary Outcome: Percentage of Participants With Early Drop Off (Prior to Completion of Cycle 3)
Description: Percent (and 95% confidence interval) of subjects who discontinue Ruxolitinib prior to completion of cycle 3
Time Frame: up to the end of cycle 3 (12 weeks)
Population: Enrolled subjects who received at least one dose of Ruxolitinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants | 16 [7.3 to 30]

8. Secondary Outcome: Percentage of Participants Who Reach Cycle 7
Description: Report percent (and 95% confidence interval) of subjects who start cycle 7(complete cycle 6)
Time Frame: Start of cycle 7
Population: Enrolled subjects who received at least one dose of Ruxolitinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants | 65 [50 to 78]

9. Secondary Outcome: Percentage of Participants With Early Drop Off (After Completion of Cycle 3 and Prior to Completion of Cycle 6)
Description: Percent (and 95% confidence interval) of subjects who discontinue after completion of 3 cycles but prior to completion of 6 cycles
Time Frame: Between cycle 3 and cycle 6
Population: Enrolled subjects who received at least one dose of Ruxolitinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants | 18 [8.8 to 32]

10. Secondary Outcome: Maximum Clinical Responses
Description: Percent (and 95% confidence interval) of subjects' maximum or "best" protocol-defined response [CR > PR > SD > PD]. Protocol-defined Response combines changes in white blood cell count, absolute neutrophil count, marrow findings and spleen size to define response (attached protocol, Section 10.6, Clinical Response, Table 6 and Table).
  Duration of maximum response was not available from the final data set. PR requires > 50% reduction in white blood cell and absolute neutrophil counts, > 50% reduction in granulocytic hyperplasia (CNL) or granulocytic dyspoiesis (aCML), and > 25% reduction in spleen size.
Time Frame: Up to 6 weeks after last dose of ruxolitinib phosphate
Population: All enrolled subjects who received at least one dose of ruxolitinib. Subject who withdraw prior to disease response evaluation are considered non-responders (PD). One subject who was inevaluable for response was included in the denominator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
percentage of participants
  Complete Response (CR) | 8 [2.3 to 20]
  Partial Response (PR) | 24 [13 to 39]
  Stable Disease (SD) | 29 [17 to 43]
  Progressive Disease (PD) | 37 [23 to 52]

11. Secondary Outcome: Change in Spleen Size, Evaluated by Ultrasound
Description: Change in spleen size (median, range) evaluated by ultrasound at the start of cycle 7 (day 1, cycle 7) and the start of study (day 1, cycle 1). Spleen volume is calculated by the conventional prolate ellipsoid method. Measure spleen width, thickness and maximum length in centimeters. Multiply width by thickness by max length by 0.524 to get the total spleen volume in cm^3. Spleen size is only one component of protocol-defined response and cannot be used to independently assess response. (see section 10.6, Clinical Response, Table 6 of attached study protocol) Change in spleen size is the difference between measurements: value at Day 1 Cycle 7 minus the value at Day 1 Cycle 1.
Time Frame: Measured on Day1 Cycle 1 and Day 1 Cycle 7
Population: Enrolled subjects receiving at least one dose of Ruxolitinib, completed 6 cycles of study drug and a had 3-dimensional spleen measurements at baseline and the start of cycle 7.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 32
cm^3 | -219.7 [-1553.8 to 1061.4]

12. Secondary Outcome: Change in Symptom Score as Measured by a Modified Myeloproliferative Neoplasm Symptom Assessment Form [MPN-SAF]
Description: Myeloproliferative Neoplasm Symptom Assessment Form Total symptom score (MPN-SAF TSS) ranges from 0 (no symptoms) to 10 (worst imaginable symptoms). The score is a sum of 10 independent measurements, generating a final score ranging from 0 - 100 and collected at baseline and on day 1, cycle 7. Change in total symptom score (TSS Median, range) is reported for those achieving day 1, cycle 7 AND responding to all 10 survey questions at baseline and Day 1, Cycle 7. Change in TSS is calculated as score on Day 1 Cycle 7 minus score at baseline.
Time Frame: Measured at baseline and Day 1 Cycle 7
Population: Enrolled subjects who received at least one dose of Ruxolitinib, completed 6 cycles of study drug and responded to all 10 survey questions at baseline and start of cycle 7.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 28
score on a scale | -3.0 [-37.0 to 8.0]

13. Secondary Outcome: Overall Survival in All Enrolled Patients
Description: Kaplan-Meier methods will be used to estimate overall survival for all enrolled patients receiving at least one dose of Ruxolitinib.
Time Frame: At stem-cell transplantation or up to 5 years after enrollment in the study
Population: Enrolled subjects receiving at least one dose of Ruxolitinib except 9 subjects who were censored at the time of stem-cell transplant
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 49
months | 17.9 [14 to NA] — Early censoring prevented estimation of upper confidence limit. We chose to censor these subjects as the increased risk associated with transplantation would otherwise contaminate the survival data.

14. Secondary Outcome: Percentage of Patients Who Achieve Clinical Response of Partial Response or Better by CSF3R Mutation Status
Description: Compute the percent (and 95% confidence interval) of patients with protocol-defined objective response (CR+PR) and IWG-defined objective response (CR+PR) at the start of cycle 7 among all enrolled patients (n = 49). Protocol-defined Response combines changes in white blood cell count, absolute neutrophil count, marrow findings and spleen size to define response (attached protocol, Section 10.6, Clinical Response, Table 6 and Table). IWG-defined Response evaluates bone marrow cellularity and myeloblast percent, absence of osteopmyelofibrosis, peripheral blood elements (white blood cell, Neutrophil, Monocyte and platelet counts, hemoglobin density, percent blasts and Neutrophil precursors), symptom resolution, dysplasia, and spleen size to determine response (attached reference). Patients who withdraw prior to the start of cycle 7 are considered non-responders.
Time Frame: Start of cycle 7
Population: All enrolled patients receiving at least one dose ruxolitinib and are evaluated for response at the start of cycle 7. Patients who withdraw prior to the start of cycle 7 are considered non-responders. One wildtype CSF3R patient was deemed inevaluable for response and was excluded from response evaluation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Wildtype CSF3R: Subjects with wildtype CSF3R
Arm/Group | Wildtype CSF3R | Mutant CSF3R
Number analyzed (Participants) | 22 | 26
percentage of participants
  Protocol-defined Response | 9 [1.1 to 29] | 54 [33 to 73]
  IWG-defined Response | 0 [0 to 0] | 15 [4.4 to 35]
Statistical Analysis 1: Comparison: Wildtype CSF3R vs Mutant CSF3R; 2-sample test for equality of proportions with continuity correction (Pearson's chi-square test statistic) comparing Wildtype and Mutant CSF3R status for protocol-defined objective response; Test type: Equivalence — 2-sample test for equality of proportions with continuity correction (Pearson's chi-square test statistic); p = 0.003, Chi-squared, Corrected — p-value for protocol-defined objective response
Statistical Analysis 2: Comparison: Wildtype CSF3R vs Mutant CSF3R; 2-sample test for equality of proportions with continuity correction (Pearson's chi-square test statistic) comparing Wildtype and Mutant CSF3R status for IWG-defined objective response; Test type: Equivalence — 2-sample test for equality of proportions with continuity correction (Pearson's chi-square); p = 0.1, Fisher Exact — p-value for IWG-defined objective response = 0.1

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected from first dose of ruxolitinib until 30 days after last dose. Any AEs occurring more than 30 days after the last dose of study drug and believed related to study drug were reported. Study drug was administered up to 96 weeks. Patients receiving ongoing clinical benefit were eligible to continue receiving study drug (up to 5 years).
Arm/Group | Treatment (Ruxolitinib Phosphate)
All-Cause Mortality (participants affected / at risk) | 36/49
Serious Adverse Events (participants affected / at risk) | 30/49
Other Adverse Events (participants affected / at risk) | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ruxolitinib Phosphate) (N=49)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood and lymphatic system disorders - Other, Specify (Blood and lymphatic system disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, Specify (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal disorders - Other, Specify (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Heart failure (Cardiac disorders) | 4 (4)
Hematoma (Vascular disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, Specify (Infections and infestations) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 6 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (6)
Urinary tract infection (Infections and infestations) | 2 (4)
Uveitis (Eye disorders) | 1 (1)
Vascular disorders - Other, Specify (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ruxolitinib Phosphate) (N=49)
Anemia (Blood and lymphatic system disorders) | 16 (28)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5)
Lymphocyte count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 7 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02092324/Prot_SAP_000.pdf